CLINICAL TRIAL: NCT00446056
Title: Montelukast, on Pediatric Bronchial Asthma in Multicenter Comparative Double-Blind Clinical Study (Phase IV) With Ketotifen Fumarate
Brief Title: Montelukast Post-Marketing Comparative Study With Ketotifen (0476-379)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-379; 2007_010
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Duration of Therapy

INTERVENTIONS:
Drug: MK0476, montelukast sodium / Duration of Treatment: 4 Weeks
Drug: Comparator: ketotifen / Duration of Treatment: 4 Weeks

SUMMARY:
The clinical study evaluates the safety of montelukast and compares montelukast to ketotifen, used as a control drug, in terms of improvement in morning peak expiratory flow (am pef) over first 2 weeks in patients with pediatric bronchial asthma aged 6 to < 15.

The effect of body weight on the efficacy and safety of montelukast will also be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Intermittent asthma, mild persistent asthma, moderate persistent asthma, or severe persistent asthma patients with 2 or more mild or moderate attacks at baseline

Exclusion Criteria:

* Patient using anti-asthma treatment or therapy including corticosteroids or oral anti-allergic drugs
* Patient with complications that will impair the judgment of efficacy of this drug
* Patient with convulsive disorders such as epilepsy or such a history
* Patient with liver disease, renal impairment, heart disease or such other complication

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 188 (Actual)
Dates: Start 2003-09-25 (Actual); Primary Completion 2004-06-16 (Actual); Study Completion 2004-06-16 (Actual)

PRIMARY OUTCOMES:
Improvement of morning peak expiratory flow over first 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Sankei N, Kenshi F, Susumu F, Shigemi Y. Cysteinyl leukotriene receptor 1 antagonist; monterukast on childhood bronchial asthma in multicenter comparative double-blind study (Phase IV) with ketotifen fumarate. J Clin Therapeut Med. 2005;21(6):605-636